CLINICAL TRIAL: NCT02164773
Title: Addition of Magnesium Sulfate to Caudal for Prevention of Emergence Agitation in Children
Brief Title: Addition of Magnesium Sulfate to Caudal to Prevent Postoperative Emergence Agitation.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Elsayed Elagamy, ashraf elagamy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: use of magnesium sulfate
Record Dates: First submitted 2014-06-03; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Agitation; Pediatric Disorder
Keywords: sevoflurane; pediatric; lower abdominal surgery; caudal; magnesium sulfate; Magnesium Sulfate Causing Adverse Effects in Therapeutic Use; Agitation States as Acute Reaction to Exceptional Stress
MeSH Terms: conditions — Psychomotor Agitation | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- magnesium sulfate (Active Comparator): magnesium sulfate 50mg caudal 1ml(5%) prepared after addition of 9ml of 0.9%normal saline to 1ml of 500mg(50%)of magnesium sulfate to be added to 1ml/kg of 0.25%of bupivacaine in caudal block in children undergoing lower abdominal surgery under sevoflurane anesthesia to prevent emergence agitation.
  Interventions: Drug: Magnesium Sulfate
- o.9%normal saline (Placebo Comparator): 0.9% of normal saline added to the conventional 0.25% bupivacaine in caudal block.
  Interventions: Drug: 0.9%normal saline

INTERVENTIONS:
Drug: Magnesium Sulfate — use of 50mg magnesium sulfate in caudal analgesia added to 1ml/kg of 0.25% of bupivacaine in children undergoing lower abdominal surgery for prevention of postoperative emergence agitation.
  Arms: magnesium sulfate
Drug: 0.9%normal saline — use of 1ml of 0.9%normal saline added to 1ml/kg of 0.25% of bupivacaine in the caudal block as placebo to compare with active comparator.
  Arms: o.9%normal saline

SUMMARY:
Emergence agitation after sevoflurane anesthesia is still a problem needed to be solved.The aim of the study is to delineate the effect of caudal magnesium sulfate in children undergoing lower abdominal surgery to prevent postoperative emergence agitation.

DETAILED DESCRIPTION:
Emergency agitation is considered one of the postoperative complication after sevoflurane anesthesia.In the enrollment of this study,children undergoing lower abdominal surgery will be enrolled in one of two groups.BM group, receive caudal magnesium sulfate 50 mg beside the conventional bupivacaine in the caudal space in ,B group, addition of 1 ml of normal saline0.9% to bupivacine .Monitoring of the postoperative emergence agitation by different emergence agitation scores with monitoring of sedation score.Detection of expected postoperative complications as nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing lower abdominal surgery for hernia repair/orchiopexy in Ain Shams University ASA physical status I under sevoflurane anesthesia.
* age from 1-6 years.

Exclusion Criteria:

* children with developmental delay
* neurological disorder.
* psychological disorder
* difficult airway
* hyperactive airway disease
* contraindication to caudal block(sacral abnormality,bleeding disorder).

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
measure of postoperative pediatric anesthesia emergence delirium PAED score | first 30 minutes postoperative
  measurement of PAED score every 5 minutes in the first 30 minutes after lower abdominal surgery in children 1-6 year age after sevoflurane anesthesia.

SECONDARY OUTCOMES:
measure of postoperative sedation score. | the first 30 minutes postoperatively
  use of sedation score as a measure of postoperative sedation expected after caudal magnesium sulfate every 5 minutes for 30 minutes after end of surgery.

OTHER OUTCOMES:
postoperative rescue propofol intravenous 1mg/kg in cases if agitation | first 30 minutes postoperative
  if emergence agitation occur giving of 1mg/kg of intravenous propofol as rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Elkateb, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Saadawy I, Boker A, Elshahawy MA, Almazrooa A, Melibary S, Abdellatif AA, Afifi W. Effect of dexmedetomidine on the characteristics of bupivacaine in a caudal block in pediatrics. Acta Anaesthesiol Scand. 2009 Feb;53(2):251-6. doi: 10.1111/j.1399-6576.2008.01818.x. Epub 2008 Dec 6. PMID 19076110
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20833531